CLINICAL TRIAL: NCT04617340
Title: The Effect of a trAnSitional Pharmacist Intervention in geRiatric Inpatients on Hospitals Visits After dischargE (ASPIRE): a Randomized Controlled Trial
Brief Title: Effect of a trAnSitional Pharmacist Intervention in geRiatric Inpatients on Hospitals Visits After dischargE
Acronym: ASPIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: S64758
Record Dates: First submitted 2020-10-29; First posted 2020-11-05 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Drug-Related Side Effects and Adverse Reactions
Keywords: Older patients; Inappropriate prescribing; Clinical pharmacy
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual care group (No Intervention): No pharmacist will be actively involved in the medication review, counseling or discharge and post-discharge procedure. In both groups the best possible preadmission drug list will be compiled for inpatients within 72 hours after admission to the geriatric ward. If potentially dangerous or life-threatening drug errors are observed in the usual care group, this will be communicated to the treating physician
- Intervention group (Experimental): The clinical pharmacist-collaborative service in the intervention group comprises six steps based on the clinical pharmacy intervention proposal of Van der Linden et al (Drugs Aging 2020).
  The first three steps focus on optimizing the drug therapy of geriatric inpatients. The remaining steps target a safe transition from the hospital to the community.
  Interventions: Other: Multifaceted clinical pharmacy intervention

INTERVENTIONS:
Other: Multifaceted clinical pharmacy intervention — 1. Assessing patient and caregiver preferences
  2. Medication reconciliation on admission
  3. Performing a comprehensive medication review before discharge
  4. Promoting safe transition
  4.a. Compiling a patient friendly medication list
  4.b.Optimizing communication with healthcare providers in primary care:
  4.b.i.Providing a copy of the medication list for the community pharmacist
  4.b.ii. Contacting the general practitioner by phone
  4.b.iii. Contacting, if applicable the home care nurse or the nurse from the nursing home by phone.
  5.A motivation interview will take place before discharge with patients and caregivers
  6.Post-discharge follow-up: 6.a.Follow-up call to discuss potential drug therapy issues, therapy adherence and to resolve any pending issues 6.b.A telepharmacology service will be provided to primary healthcare professionals as a means to consult the ward-based clinical pharmacists and/or research team after discharge.
  Arms: Intervention group

SUMMARY:
A randomized controlled trial will be performed in geriatric inpatients to investigate the impact of a multifaceted clinical pharmacy intervention on health related outcomes.

DETAILED DESCRIPTION:
Since drug-related harm remains persistently prevalent in older adults, there is an urgent and unmet clinical need to optimize pharmacotherapy both during hospital stay and after discharge Therefore, we aim to perform a randomized controlled trial in geriatric inpatients to investigate the impact of a multifaceted clinical pharmacy intervention on health related outcomes. The primary objective is to reduce all-cause unplanned hospital visits in geriatric inpatients. Secondary objective are to optimize drug therapy in geriatric inpatients and improve their health; To empower and educate patients, caregivers,community pharmacists and physicians regarding drug regimen decisions to maximize therapy adherence and the understanding of the (de)prescribing process and to enhance healthy ageing; To optimize transitional care from the hospital to primary care.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to one of the study wards under supervision of a geriatrician
* A written informed consent by the patient or his/her representative
* Discharged from the hospital

Exclusion Criteria:

* Admitted for a maximum of one day
* Unable to understand Dutch
* Being in a palliative stage as stated in their medical record with active withdrawal of drug therapy
* Patients being discharged to another ward within the same hospital or to another hospital

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 827 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-09-27 (Actual)

PRIMARY OUTCOMES:
Time to all-cause unplanned hospital visit after discharge. | up to six months after discharge
  An unplanned hospital visit is defined as an unplanned hospital admission or an emergency department visit

SECONDARY OUTCOMES:
General practitioners contacts | Up to six months after discharge
  Number of general practitioners contacts
Mortality | Up to six months after discharge
  Death date
Other types of hospital visits | Up to six months after discharge
  Number of planned hospital admissions, number of emergency department visits, number of unplanned hospital admissions
Drug-related readmissions | Up to six months after discharge
  Number of drug related readmissions
Fall incidents | Up to one month after discharge
  Number of falls
Patient reported drug related problems | Up to one month after discharge
  Number of drug related problems
Change in Quality of life | on admission, one month after discharge and six months after discharge
  five-level version of the EuroQol five-dimensional (EQ5D) descriptive system (EQ-5D-5L) questionnaire. values will be tranformed using a value set to a score from 0 - 1 (a higher score indicating a better quality of life)
Differences in pain | Up to one month after discharge
  Numeric Rating Scale (NRS score) once a week (min 0 - max 10), a higher score indicating more pain
Medications | On admission, at discharge and one month after discharge
  Number of medications
Medication adherence | On admission and one month after discharge
  BAASIS tool
Potentially inappropriate medications | On admission, at discharge and one month after discharge
  RASP tool
Cost-effectiveness | Up to six months after discharge
  Healthcare related costs and Medicine productivity costs

CONTACTS AND LOCATIONS:
Overall Officials: Jos Tournoy, prof, Principal Investigator — Department of Public Health and Primary care, KU Leuven, Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No
IPD will not be made available publicly due to privacy or ethical restrictions, but data that support the findings of this study will be available upon reasonable request

REFERENCES:
- [Background] Van der Linden L, Hias J, Walgraeve K, Flamaing J, Tournoy J, Spriet I. Clinical Pharmacy Services in Older Inpatients: An Evidence-Based Review. Drugs Aging. 2020 Mar;37(3):161-174. doi: 10.1007/s40266-019-00733-1. PMID 31919802
- [Derived] Hellemans L, Blocquiaux L, Hias J, Walgraeve K, Liesenborghs A, Lammens A, Deschodt M, Tournoy J, Van der Linden L. Effect of a Multifaceted Pharmacist-Led Intervention on Medication Appropriateness and Medication Burden in Patients Admitted to an Acute Geriatric Ward: Results from the ASPIRE Trial. Drugs Aging. 2026 Jan 31. doi: 10.1007/s40266-026-01278-w. Online ahead of print. PMID 41619153
- [Derived] Hias J, Hellemans L, Laenen A, Walgraeve K, Liesenborghs A, De Geest S, Luyten J, Spriet I, Flamaing J, Van der Linden L, Tournoy J. The effect of a trAnSitional Pharmacist Intervention in geRiatric inpatients on hospital visits after dischargE (ASPIRE): Protocol for a randomized controlled trial. Contemp Clin Trials. 2022 Aug;119:106853. doi: 10.1016/j.cct.2022.106853. Epub 2022 Jul 14. PMID 35842106